CLINICAL TRIAL: NCT04329494
Title: Safety and Efficacy of Pressurized Intraperitoneal Aerosolized Chemotherapy (PIPAC) in Ovarian, Uterine, Appendiceal, Colorectal, and Gastric Cancer Patients With Peritoneal Carcinomatosis (PC)
Brief Title: PIPAC for the Treatment of Peritoneal Carcinomatosis in Patients With Ovarian, Uterine, Appendiceal, Colorectal, or Gastric Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19184; NCI-2020-01254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19184 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-03-13; First posted 2020-04-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVB Gastric Cancer AJCC v8; Malignant Uterine Neoplasm; Metastatic Appendix Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Gastric Carcinoma; Metastatic Malignant Neoplasm in the Peritoneum; Metastatic Malignant Solid Neoplasm; Metastatic Ovarian Carcinoma; Pathologic Stage IV Gastric Cancer AJCC v8; Peritoneal Carcinomatosis; Postneoadjuvant Therapy Stage IV Gastric Cancer AJCC v8; Stage IV Appendix Carcinoma AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Uterine Corpus Cancer AJCC v8; Stage IVA Appendix Carcinoma AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Uterine Corpus Cancer AJCC v8; Stage IVB Appendix Carcinoma AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Uterine Corpus Cancer AJCC v8; Stage IVC Appendix Carcinoma AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Uterine Neoplasms; Appendiceal Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms; Peritoneal Neoplasms | interventions — Biopsy; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Doxorubicin; Fluorouracil; dehydroftorafur; Hyperthermic Intraperitoneal Chemotherapy; Irinotecan; Leucovorin; Mitomycin; Mitozytrex; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Arm I (PIPAC, doxorubicin, cisplatin) - Not recruiting (Experimental): Patients with ovarian, uterine, or gastric cancer, undergo PIPAC with doxorubicin IP, followed by cisplatin IP. Treatment repeats every 4-6 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Drug: Cisplatin; Drug: Doxorubicin; Device: Intraperitoneal Chemotherapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (PIPAC, oxaliplatin, leucovorin, fluorouracil) - Not recruiting (Experimental): Patients with colorectal or appendiceal cancer undergo PIPAC with oxaliplatin IP. For cycles 2 and 3, patients receive leucovorin IV over 10 minutes and fluorouracil IV over 15 minutes 1-24 hours before undergoing PIPAC. Treatment repeats every 4-6 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Drug: Fluorouracil; Device: Intraperitoneal Chemotherapy; Drug: Leucovorin; Drug: Oxaliplatin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (PIPAC, mitomycin, FOLFIRI) - Not recruiting (Experimental): Patients with colorectal or appendiceal cancer who have undergo at least 4 months (or 8 cycles) of first-line standard of care chemotherapy but have not progressed on second line chemotherapy undergo PIPAC with mitomycin IP. Patients also receive standard of care irinotecan IV over 90 on day 1, leucovorin IV over 30 minutes on day 1, and fluorouracil IV on days 1-2 during weeks 2, 4, 8, 10, 14 and 16. Treatment repeats every 4-6 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Drug: Fluorouracil; Device: Intraperitoneal Chemotherapy; Drug: Irinotecan; Drug: Leucovorin; Drug: Mitomycin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm IV (PIPAC, Cisplatin and nab-paclitaxel) (Experimental): Patients with recurrent ovarian cancer ( platinum-resistent or platinum metastases) patients with unresectable peritoneal metastases who are not candidates for cytoreductive surgery, at least 6 months after completion of first-line standard of care chemotherapy, and no bowel obstruction. Treatment for each 28-day cycle will consist of PIPAC with cisplatin (15 mg/m2) and nab-paclitaxel (90 mg/m2) on D1 every 28 days. A dose de-escalation plan is provided if the starting dose is not well-tolerated.
  Interventions: Procedure: Biopsy; Drug: Cisplatin; Device: Intraperitoneal Chemotherapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Drug: Cisplatin — Given via PIPAC
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm I (PIPAC, doxorubicin, cisplatin) - Not recruiting; Arm IV (PIPAC, Cisplatin and nab-paclitaxel)
Drug: Doxorubicin — Given via PIPAC
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Arm I (PIPAC, doxorubicin, cisplatin) - Not recruiting
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm II (PIPAC, oxaliplatin, leucovorin, fluorouracil) - Not recruiting; Arm III (PIPAC, mitomycin, FOLFIRI) - Not recruiting
Device: Intraperitoneal Chemotherapy — Undergo PIPAC
  Other Names: Intraperitoneal Therapy
Drug: Irinotecan — Given IV
  Arms: Arm III (PIPAC, mitomycin, FOLFIRI) - Not recruiting
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
  Arms: Arm II (PIPAC, oxaliplatin, leucovorin, fluorouracil) - Not recruiting; Arm III (PIPAC, mitomycin, FOLFIRI) - Not recruiting
Drug: Mitomycin — Given via PIPAC
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
  Arms: Arm III (PIPAC, mitomycin, FOLFIRI) - Not recruiting
Drug: Oxaliplatin — Given via PIPAC
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
  Arms: Arm II (PIPAC, oxaliplatin, leucovorin, fluorouracil) - Not recruiting
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects of pressurized intraperitoneal aerosol chemotherapy (PIPAC) in treating patients with ovarian, uterine, appendiceal, stomach (gastric), or colorectal cancer that has spread to the lining of the abdominal cavity (peritoneal carcinomatosis). Chemotherapy drugs, such as cisplatin, doxorubicin, oxaliplatin, leucovorin, fluorouracil, mitomycin, and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. PIPAC is a minimally invasive procedure that involves the administration of intraperitoneal chemotherapy. The study device consists of a nebulizer (a device that turns liquids into a fine mist), which is connected to a high-pressure injector, and inserted into the abdomen (part of the body that contains the digestive organs) during a laparoscopic procedure (a surgery using small incisions to introduce air and to insert a camera and other instruments in the abdominal cavity for diagnosis and/or to perform routine surgical procedures). Pressurization of the liquid chemotherapy through the study device results in aerosolization (a fine mist or spray) of the chemotherapy intra-abdominally (into the abdomen). Giving chemotherapy through PIPAC may reduce the amount of chemotherapy needed to achieve acceptable drug concentration, and therefore potentially reduces side effects and toxicities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of pressurized intraperitoneal aerosol chemotherapy (PIPAC) in 3 groups of patients: peritoneal carcinomatosis (PC) due to primary ovarian, uterine, or gastric carcinoma (Arm 1); PC due to primary colorectal or appendiceal carcinoma (Arm 2).

II. To evaluate safety of PIPAC and identify the maximum tolerated dose (MTD) of PIPAC with MMC in patients with PC due to colorectal or appendiceal carcinoma (Arm 3).

SECONDARY OBJECTIVES:

I. Ability to proceed to cytoreduction with/without hyperthermic intraperitoneal chemotherapy (HIPEC) (Arm 3 patients).

II. Efficacy will be assessed by:

Ia. Response Evaluation Criteria in Solid Tumors (RECIST), if available, version 1.1 via computed tomography (CT) scan at baseline (week 10, and 6 weeks after completing treatment; and at 18 weeks).

Ib. Peritoneal regression grading score (PRGS) via biopsy at each cycle (both pre-PIPAC and post-PIPAC peritoneal samples will be obtained).

Ic. Peritoneal carcinomatosis index (PCI) at the time of laparoscopy. II. Post-operative surgical complications by Claven-Dindo classification evaluated at 4, 10, and 16 weeks (4 weeks after each PIPAC).

III. Progression-free survival. IV. PIPAC technical failure rate. V. Patient-reported health state/quality of life and symptoms before treatment and at 6, 12, and 18 weeks as measured by the European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ-5D-5L) and MD Anderson Symptom Inventory (MDASI).

VI. Functional status, as measured by the number of daily steps before and after treatments (Vivofit 4 wristband pedometer - Garmin Company).

EXPLORATORY OBJECTIVE:

I. Correlative/translational studies to characterize the tumor microenvironment, subclonal evolution, genomics, and pharmacokinetics of peritoneal tumors.

OUTLINE: Patients are assigned to 1 of 3 arms.

ARM I: Patients with ovarian, uterine, or gastric cancer, undergo PIPAC with doxorubicin intraperitoneally (IP), followed by cisplatin IP. Treatment repeats every 4-6 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients with colorectal or appendiceal cancer undergo PIPAC with oxaliplatin IP. For cycles 2 and 3, patients receive leucovorin intravenously (IV) over 10 minutes and fluorouracil IV over 15 minutes 1-24 hours before undergoing PIPAC. Treatment repeats every 4-6 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

ARM III: Patients with colorectal or appendiceal cancer who have undergo at least 4 months (or 8 cycles) of first-line standard of care chemotherapy but have not progressed on second line chemotherapy undergo PIPAC with mitomycin IP. Patients also receive standard of care irinotecan IV over 90 on day 1, leucovorin IV over 30 minutes on day 1, and fluorouracil IV on days 1-2 during weeks 2, 4, 8, 10, 14 and 16. Treatment repeats every 4-6 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Patients must have histologically confirmed ovarian, uterine, gastric, appendiceal or colorectal cancer with PC
* Prior IP chemotherapy is permitted
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9 g/dl
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) and aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x ULN, unless liver metastases (Arm 1) are present or unless patients is know to have chronic liver disease (hepatitis) in which case AST and ALT must be =< 5 x ULN
* Alkaline phosphatase =< 2 x ULN
* Serum creatinine (sCr) =< 1.5 x ULN, or creatinine clearance (Ccr) >= 40 ml/min as calculated by the Cockcroft-Gault formula
* No contraindications for a laparoscopy
* The peritoneal disease does not have to be measurable by RECIST 1.1 but needs to be visible on cross sectional imaging or diagnostic laparoscopy
* Patients must have progressed on at least one evidence-based chemotherapeutic regimen (Arm 1 and 2). For Arm 3, patients should have stable or responsive disease on at least 4 months first-line systemic chemotherapy
* For patients with a known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Women of childbearing potential (WOCBP) and male patients with WOCBP partner must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Post menopause is define as:

  * Amenorrhea >= 12 consecutive months without another cause or
  * For women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
  * Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential
* INCLUSION TO PROCEED WITH PIPAC: Laparoscopy findings must meet all of the below criteria in order to proceed to PIPAC:

  * PIPAC access is feasible
  * There is room for aerosol therapy
  * There is no evidence of impending bowel obstruction
  * =< 5 L of ascites
  * Not a candidate for cytoreduction and HIPEC

Exclusion Criteria:

* Gastric and colorectal/appendiceal:

  * Extra-peritoneal metastatic disease
* Arm 1 (ovarian, uterine, gastric): Previous treatment with maximum cumulative doses of doxorubicin, daunorubicin, epirubicin, idarubicin, and/or other anthracyclines and anthracenediones
* Arm 2 (colorectal/appendiceal): Known dihydropyrimidine dehydrogenase deficiency (DPD) deficiency
* Arm 2 (colorectal/appendiceal): Bowel obstruction requiring nasogastric tube, percutaneous endoscopic gastrostomy or exclusive total parenteral nutrition
* Arm 2 (colorectal/appendiceal): Prior unanticipated severe reaction or hypersensitivity to platinum based compounds
* Arm 2 (colorectal/appendiceal): Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1), with the exception of alopecia, hearing loss, or non-clinically significant laboratory abnormalities. Grade 2 peripheral neuropathy is permitted
* Arm 2 (colorectal/appendiceal): Life expectancy of less than 6 months
* Arm 2 (colorectal/appendiceal): Chemotherapy or surgery within the last 4 weeks prior to enrollment (6 weeks for prior bevacizumab therapy). Five half-lives for other anti-cancer agents
* Arm 2 (colorectal/appendiceal): Previous anaphylactic reaction to the chemotherapy drug used
* Arm 2 (colorectal/appendiceal): Patients may not be receiving any other investigational or concurrent anti-cancer agents
* Arm 2 (colorectal/appendiceal): Ascites due to decompensated liver cirrhosis; portal vein thrombosis
* Arm 2 (colorectal/appendiceal): Simultaneous tumor debulking with gastrointestinal resection
* Arm 2 (colorectal/appendiceal): Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, severe myocardial insufficiency, recent myocardial infarction, severe arrhythmias, severe renal impairment, myelosuppression, or severe hepatic impairment
* Arm 2 (colorectal/appendiceal): Immunocompromised patients such as those with an immunosuppressive medication or a known disease of the immune system
* Arm 2 (colorectal/appendiceal): Involvement in the planning and conduct of the study
* Arm 2 (colorectal/appendiceal): Pregnancy
* Arm 2 (colorectal/appendiceal): Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Arm 2 (colorectal/appendiceal): New York Heart Association (NYHA) class 3 or 4; myocardial infarction, acute coronary syndrome, diabetes mellitus with ketoacidosis or chronic obstructive pulmonary disease (COPD) requiring hospitalization in the preceding 6 months
* Arm 2 (colorectal/appendiceal): Major systemic infection requiring antibiotics 72 hours or less prior to the first dose of study drug
* Arm 2 (colorectal/appendiceal): Exclusive total parenteral nutrition
* Arm 2 (colorectal/appendiceal): Prior intra-abdominal aerosol chemotherapy
* Arm 3 (colorectal/appendiceal): Progression on first- AND second-line systemic therapy
* Arm 3 (colorectal/appendiceal): Hematologic toxicities requiring significant dose reductions while on systemic chemotherapy
* Arm 3 (colorectal/appendiceal): Intolerance to prior 5-FU at 2400mg/m^2 IV every 2 weeks or to irinotecan at 180mg/m^2. Intolerance is defined as the need of significant dose reduction or treatment interruption of > 1 week due to toxicity
* Arm 3 (colorectal/appendiceal): Known DPD deficiency
* Arm 3 (colorectal/appendiceal): Bowel obstruction requiring nasogastric tube, percutaneous endoscopic gastrostomy or exclusive total parenteral nutrition
* Arm 3 (colorectal/appendiceal): Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1), with the exception of alopecia, hearing loss, or non-clinically significant laboratory abnormalities. Grade 2 peripheral neuropathy is permitted
* Arm 3 (colorectal/appendiceal): Life expectancy of less than 6 months
* Arm 3 (colorectal/appendiceal): Chemotherapy or surgery within the last 2 weeks prior to enrollment (6 weeks for prior bevacizumab therapy). Five half-lives for other anti-cancer agents
* Arm 3 (colorectal/appendiceal): Previous anaphylactic reaction to the chemotherapy drug used
* Arm 3 (colorectal/appendiceal): Patients may not be receiving any other investigational anti-cancer agents
* Arm 3 (colorectal/appendiceal): Ascites due to decompensated liver cirrhosis; portal vein thrombosis
* Arm 3 (colorectal/appendiceal): Simultaneous tumor debulking with gastrointestinal resection
* Arm 3 (colorectal/appendiceal): Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, severe myocardial insufficiency, recent myocardial infarction, severe arrhythmias, severe renal impairment, myelosuppression, or severe hepatic impairment
* Arm 3 (colorectal/appendiceal): Immunocompromised patients such as those with an immunosuppressive medication or a known disease of the immune system
* Arm 3 (colorectal/appendiceal): Involvement in the planning and conduct of the study
* Arm 3 (colorectal/appendiceal): Pregnancy
* Arm 3 (colorectal/appendiceal): Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Arm 3 (colorectal/appendiceal): New York Heart Association (NYHA) class 3 or 4; myocardial infarction, acute coronary syndrome, diabetes mellitus with ketoacidosis or chronic obstructive pulmonary disease (COPD) requiring hospitalization in the preceding 6 months
* Arm 3 (colorectal/appendiceal): Major systemic infection requiring antibiotics 72 hours or less prior to the first dose of study drug
* Arm 3 (colorectal/appendiceal): Exclusive total parenteral nutrition
* Arm 3 (colorectal/appendiceal): Prior intra-abdominal aerosol chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2028-01-05 (Estimated); Study Completion 2028-01-05 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities | Up to 18 weeks
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Summarized by type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment, and reversibility or outcome.
Incidence of adverse events | From day 1 of protocol therapy until week 18
  Assessed using CTCAE v.5.0. Summarized by grade and attribution. Post-surgical complications will be assessed by Clavien-Dindo classification.

SECONDARY OUTCOMES:
Percentage of evaluable patients who have achieved complete response (CR), partial response (PR), or stable disease (SD) | At baseline, following the second cycle (week 10), and 6 weeks after completing treatment (at 18 weeks/off-study)
  Assessed by Response Evaluation Criteria in Solid Tumors criteria version 1.1 via computed tomography (CT) scan. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach by Clopper and Pearson.
Percentage of evaluable patients who have achieved CR, PR, or SD | At the time of laparoscopy (or CT imaging if laparoscopy is not planned during surgery)
  Assessed by Peritoneal Carcinomatosis Index. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach by Clopper and Pearson.
Percentage of evaluable patients who have achieved a decrease in Peritoneal Regression Grading Score over successive biopsies | Up to 18 weeks
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach by Clopper and Pearson.
Progression-free survival | Time from first pressurized intraperitoneal aerosolized chemotherapy (PIPAC) procedure, assessed up to 1 year
  Described using the Kaplan-Meier method.
Post-surgical complications | At 4 weeks after each PIPAC
  Assessed by Clavien-Dindo classification. Results will be strictly descriptive in nature.
PIPAC technical failure rate | Up to 3 years
Functional status | Up to 18 weeks
  Measured by the number of daily steps before and after treatments (Vivofit 4 wristband pedometer - Garmin Company).
Cytoreductive surgery rate (Arm 3) | Up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thanh H Dellinger, MD, Principal Investigator — City of Hope Medical Center; Mustafa Raoof, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York